CLINICAL TRIAL: NCT01486173
Title: Early Nutrition and Neurological Development of Very Preterm Infants
Acronym: EPINUTRI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lapillonne, Alexandre, M.D. (Individual)
Responsible Party: Principal Investigator, Alexandre Lapillonne, M.D., Ph.D., Professor of Pediatrics, Lapillonne, Alexandre, M.D.
Other Study IDs: 2011-mars-12551
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Infant, Premature, Diseases; Infant Nutrition Disorders; Development; Delayed, Mental
Keywords: PUFA; Iron; Neurological development; Premature infant
MeSH Terms: conditions — Infant, Premature, Diseases; Infant Nutrition Disorders; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Premature infants with a GA < 32 Weeks
- New born with a GA > 37Weeks

SUMMARY:
The main goal of this study is to determine the association between:

* the quantity of mother's milk and duration of breastfeeding
* the intake of polyunsaturated fatty acids and iron during hospitalization and the development of preterm infants born with a GA < 32 weeks.

ELIGIBILITY:
Inclusion criteria:

* infants with a gestational age < 32 weeks already included in the EPIPAGE2 study
* agreement of parents

Exclusion criteria:

* death during hospitalisation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subsample of infants born very preterm (before 32 weeks of gestation) otherwise included in the French national cohort EPIPAGE 2
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Neurological development at 2 years of age | 3 years
  Age and Stages Questionnaire at 2 years of age
  Brunet Lezine test

SECONDARY OUTCOMES:
Nutritional status at time of discharge | 1 year
  Polyunsaturated fatty acids status
  Iron status

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lapillonne, M.D., Ph.D., Study Director — Alexandre Lapillonne
Locations (1):
- Necker hospital, Paris, Île-de-France Region, France